CLINICAL TRIAL: NCT06143033
Title: A Clinical Trial to Evaluate the Effects of an Eye Serum on Improving the Appearance of the Periorbital Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dime Beauty Co. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20363
Record Dates: First submitted 2023-11-05; First posted 2023-11-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Periorbital Area

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DIME Beauty Luminosity Eye Serum (Experimental): Participants will use the serum twice daily after their morning and evening skincare routine (i.e., after cleansing, and applying facial serums and moisturizers), but before the application of sunscreen.
  Interventions: Other: DIME Beauty Luminosity Eye Serum

INTERVENTIONS:
Other: DIME Beauty Luminosity Eye Serum — Test product contains: Water/Aqua, Organic Aloe Vera Juice, Lycium Barbarum (Goji Berry) Fruit Extract, Vitis Vinifera (Grape Seed) Extract, Cucumis Sativus (Cucumber) Extract, Glycerin, Niacinamide, Squalane, Camellia Seed Oil, DL-Panthenol (Vitamin B5), Carbomer, Sodium Hyaluronate, Ammonium Acryloyldimethyltaurate/VP Copolymer, Phenoxyethenol, Caprylyl Glycol, Acacia Senegal Gum, Caffeine, Helianthus Annuus (Sunflower) Seed Oil, Malus Domestica (Apple) Fruit Stem Cell Extract, Argania Spinosa (Argan) Sprout Stem Cell Extract, Tetrahexyldecyl Ascorbate (Vitamin C), Acetyl Tetrapeptide, Acetyl Hexapeptide-8, Vitamin E Mixed Tocopherols, Sodium Hydroxide.

SUMMARY:
This study will evaluate the efficacy of the DIME Beauty Luminosity Eye Serum in improving the appearance of skin in the periorbital eye area. This study will last for 60 days. The study will be conducted as a single-arm trial in which all participants will use the test products. Participants will be required to complete questionnaires at Baseline, Day 30, and Day 60, photos will be taken at Baseline, Day 30, and Day 60, and expert skin grading will take place at Baseline and Day 60.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18-65.
* Have visible dark circles under the eyes.
* Have puffy eyes.
* Have bags under the eyes.
* Have visible fine lines and wrinkles around the eyes.
* Have a smartphone or camera to take before-and-after selfies.

Exclusion Criteria:

* Anyone not in good health.
* Anyone who has any chronic health conditions such as oncological or psychiatric disorders.
* Anyone who has any known serious allergic reactions that require the use of an Epi-Pen.
* Anyone who is pregnant, breastfeeding, or wanting to become pregnant over the next three months.
* Anyone who cannot/ will not commit to the study protocol.
* Anyone with a history of substance abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Change in appearance of periorbital puffiness. [Baseline to Day 60] | 60 days
  Measured via expert skin grading of before & after photos conducted by a board-certified dermatologist.
Change in appearance of dark circles underneath eyes. [Baseline to Day 60] | 60 days
  Measured via expert skin grading of before & after photos conducted by a board-certified dermatologist.
Change in participants' perception of the appearance of periorbital puffiness. [Baseline to Day 60] | 60 days
  Measured via study-specific surveys. Surveys will be completed by participants and are designed using a 5-point Likert scale, with th 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Change in participants' perception of the appearance of dark circles underneath eyes. [Baseline to Day 60] | 60 days
  Measured via study-specific surveys. Surveys will be completed by participants and are designed using a 5-point Likert scale, with th 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

SECONDARY OUTCOMES:
Change in appearance of fine lines and wrinkles in the eye area. [Baseline to Day 60] | 60 days
  Measured via expert skin grading of before & after photos conducted by a board-certified dermatologist.
Change in participants' perception of the appearance of fine lines and wrinkles in the eye area. [Baseline to Day 60] | 60 days
  Measured via study-specific surveys. Surveys will be completed by participants and are designed using a 5-point Likert scale, with th 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided